CLINICAL TRIAL: NCT05001503
Title: Pivotal Phase, Randomised Controlled Trial to Demonstrate a Reduction in the Number of Oliguria Events in Patients Being Managed in a Critical Care Unit, Following Cardiac Surgery, When a Novel Oliguria Prediction Tool (STABILITY UO) is Used to Identify Patients at Risk, Compared to Standard of Care.
Brief Title: Controlled Trial to Demonstrate a Reduction in the Number of Oliguria Events in Patients Being Managed in a Critical Care Unit, Following Cardiac Surgery, When a Novel Oliguria Prediction Tool (STABILITY UO) is Used to Identify Patients at Risk, Compared to Standard of Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rinicare Ltd (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Stability UO 001 v1.0
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The clinical team has access to the Stability UO software. All other care is given as standard.
  Interventions: Device: Stability UO
- Control Group (No Intervention): Standard care given.

INTERVENTIONS:
Device: Stability UO — STABILITY UO is a standalone software, based on a Bayesian model, which quantifies the risk of an individual patient developing severe oliguria (0.3mg/kg/hr for 6 hours). The model identifies at risk patients by predicting future urine output, using only previously recorded urine output values for that individual, allowing clinicians to see the predicted risk of a patient developing severe oliguria in real time.
  Arms: Intervention Group

SUMMARY:
Acute kidney injury (AKI) is experienced by 12% of patients following surgery and in up to 50% of patients following cardiac surgery. It is associated with an increased risk of death and prolonged stay in critical care after surgery. In addition to the patient impact, AKI costs the NHS alone between £434m and £620m per year.

One way that AKI is diagnosed is by looking at a patient's urine output and checking how much is produced over time. If this value is too low for a patient, they are diagnosed with oliguria. Too many of these oliguria events leads to a diagnosis of AKI. The product to be tested (Stability UO) aims to reduce the number of patients who suffer three or more oliguria events after surgery by processing the data entered by the care team and providing the care team with additional information about the patient's risk of oliguria over the next six hours.

Patients over 18 who present at Manchester University NHS Foundation Trust for non-emergency cardiac surgery will be screened and asked to consent to be randomised as part of the trial. Patients undergoing certain operations and those with unsuitable medical history (e.g. patients being treated for dialysis) will not be invited to participate. The randomisation will determine if their care team has access to the Stability UO software after surgery. While the care team looks after the patients in the cardiothoracic critical care unit (CTCCU) after surgery, they will enter that the patient's weight and amount of urine passed each hour into the software and review the output. The primary questions the study will answer is if there is a difference between number of oliguria events between the two groups of patients.

The study is funded by the device manufacturer: Rinicare Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the study, including being able to receive study materials at least 24 hours prior to their planned operation,
* Patient is Male or Female, aged 18 years or above,
* Patient is due to undergo elective or urgent cardiac surgery, and who is expected to be managed on the CTCCU postoperatively,
* In the Investigator's opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

* Patients undergoing emergency surgery (i.e surgery that has to take place in the next available theatre even if this is out of standard operating hours)
* Patients having ventricular assist device implantation,
* Patients receiving a heart transplant,
* Patients who would be unable to be treated by standard of care CTCCU therapies and practices,
* Patients who are receiving pre or intra-operative dialysis or haemofiltration.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Absolute Risk Reduction (ARR) of patients experiencing ≥3 oliguria events. | post cardiac surgery CTCCU stay (average 2-5 days with some staying more than 3 months)
  An oliguria event is defined as an hourly urine output of less than 0.5ml/kg/hr.

SECONDARY OUTCOMES:
Incidence of oliguria events during post cardiac surgery CTCCU stay | post cardiac surgery CTCCU stay (average 2-5 days with some staying more than 3 months)
  An oliguria event is defined as an hourly urine output of less than 0.5ml/kg/hr.
Absolute Risk (AR), Relative Risk (RR), Relative Risk Reduction (RRR) of severe oliguria events | post cardiac surgery CTCCU stay (average 2-5 days with some staying more than 3 months)
  An severe oliguria event is defined as an hourly urine output of less than 0.3ml/kg/hr.
Median length of total stay in hospital | post cardiac surgery CTCCU stay (average 2-5 days with some staying more than 3 months)
  median length of stay in hospital
Change in post-operative serum creatinine concentration | post cardiac surgery CTCCU stay (average 2-5 days with some staying more than 3 months)
  Standard blood test to measure serum creatinine concentration (umol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Mosca, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Wythenshawe Hospital (Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howitt SH, Oakley J, Caiado C, Goldstein M, Malagon I, McCollum C, Grant SW. A Novel Patient-Specific Model for Predicting Severe Oliguria; Development and Comparison With Kidney Disease: Improving Global Outcomes Acute Kidney Injury Classification. Crit Care Med. 2020 Jan;48(1):e18-e25. doi: 10.1097/CCM.0000000000004074. PMID 31663925
- [Background] Howitt SH, Grant SW, Caiado C, Carlson E, Kwon D, Dimarakis I, Malagon I, McCollum C. The KDIGO acute kidney injury guidelines for cardiac surgery patients in critical care: a validation study. BMC Nephrol. 2018 Jun 25;19(1):149. doi: 10.1186/s12882-018-0946-x. PMID 29940876